CLINICAL TRIAL: NCT02635191
Title: Tailored Therapy Versus Standard Triple Therapy for Helicobacter Pylori Eradication in Children: A Randomized Trial
Brief Title: Tailored Therapy for Helicobacter Pylori in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Xiwei Xu, Chief of Gastroenterology Department, Beijing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCH-HP-001
Record Dates: First submitted 2015-11-25; First posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Therapy; Children
MeSH Terms: interventions — Rabeprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored Group (Experimental): In tailored therapy, medications will be adjusted according to the antimicrobial susceptibility testing (including Clarithromycin sensitivity) and cytochrome P450 isoenzyme 2C19 genotype. 10 days regimen will be prescribed.
  Interventions: Drug: Tailored Group
- Standard group (Active Comparator): In standard triple therapy, children will be treated by Omeprazole(0.8-1.0mg/kg.d,bid), Amoxicillin (30-50mg/kg.d bid)and Clarithromycin (15-20mg/kg.d bid) for 10 days.
  Interventions: Drug: Standard group

INTERVENTIONS:
Drug: Tailored Group — All the patients who enrolled in this arm will be received endoscopy followed by biopsy for antimicrobial susceptibility testing and cytochrome P450 isoenzyme 2C19 genotype. 10 days tailored therapy will be given including one Proton Pump Inhibitor ( Rabeprazole0.4-0.5mg/kg.d,bid. or Esomeprazole0.8-1.0mg/kg.d,bid) and two antibiotics (Amoxicillin30-50mg/kg.d bid, Clarithromycin15-20mg/kg.d bid, Metronidazole15-20mg/kg.d bid ) based on the cytochrome P450 isoenzyme 2C19 genotype and the antimicrobial susceptibility.
  Other Names: "Rabeprazole"" Pariet®"; "Esomeprazole"" Nexium®"; "Metronidazole""Yabao®"; "Amoxicillin""Tongdamoxing®"
  Arms: Tailored Group
Drug: Standard group — All the patients who enrolled in this arm will be treated by Omeprazole(0.8-1.0mg/kg.d,bid), Amoxicillin (30-50mg/kg.d bid)and Clarithromycin (15-20mg/kg.d bid) .
  Other Names: "Omeprazole"" LosecMUPS®"; "Amoxicillin""Tongdamoxing®"; "Clarithromycin""Klacid®"
  Arms: Standard group

SUMMARY:
This study is designed to compare the eradication rates，safety and compliance of tailored therapy to those of standard triple therapy in children with H. pylori infection. The primary purpose is to compare the eradication rates of children with H. pylori infection treated with tailored therapy to those treated with standard triple therapy. The secondary purpose is to evaluate the safety, compliance and factors that might affect eradication rates.

DETAILED DESCRIPTION:
Between March 2014 and March 2016, 200 children with upper gastrointestinal symptoms (4-18 years) and H. pylori infection will be recruited at Beijing Children Hospital.After the informed consents are obtained from the guardians, the children will be randomly classified into the two group: 10 days standard triple therapy (Omeprazole 0.8-1.0mg/kg.d,bid, Amoxicillin 30-50mg/kg.d bid， Clarithromycin 15-20mg/kg.d bid), or 10 days tailored therapy including one Proton Pump Inhibitor ( Rabeprazole 0.4-0.5mg/kg.d,bid. or Esomeprazole 0.8-1.0mg/kg.d,bid) and two antibiotics (Amoxicillin 30-50mg/kg.d bid, Clarithromycin 15-20mg/kg.d bid, Metronidazole15-20mg/kg.d bid) based on antibiotics susceptibility and cytochrome P450 isoenzyme 2C19 genotype. Eradication status will be reassessed in four weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of H. pylori infection.
* Presence of upper gastrointestinal symptoms.
* Referred for upper endoscopy at Beijing Children's Hospital

Exclusion Criteria:

* Presence of endoscopy contraindications
* The administration of any drug that could influence the study results including proton pump inhibitors, H2-receptor blockers, bismuth salts and antibiotics within the previous four weeks;
* Gastrointestinal malignancy;
* Previous gastric or esophageal surgery;
* Severe concomitant diseases
* History of allergy to any of the study drugs;

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Compare the eradication rates in each group | One month after treatment
  The efficacy of H. pylori eradication between the standard triple therapy and tailored therapy based on the results of antimicrobial resistance(including Clarithromycin sensitivity) by using H. pylori culture and cytochrome P450 isoenzyme 2C19 genotype. Eradication status will be reassessed in one month after treatment.

OTHER OUTCOMES:
Compare the adverse reactions in each group | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Xiwei Xu, MD, Principal Investigator — Beijing Children's Hosipital of Capital Medical University,China
Locations (1):
- Beijing, China

REFERENCES:
- [Background] Liu G, Xu X, He L, Ding Z, Gu Y, Zhang J, Zhou L. Primary antibiotic resistance of Helicobacter pylori isolated from Beijing children. Helicobacter. 2011 Oct;16(5):356-62. doi: 10.1111/j.1523-5378.2011.00856.x. PMID 21923681
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Koletzko S, Jones NL, Goodman KJ, Gold B, Rowland M, Cadranel S, Chong S, Colletti RB, Casswall T, Elitsur Y, Guarner J, Kalach N, Madrazo A, Megraud F, Oderda G; H pylori Working Groups of ESPGHAN and NASPGHAN. Evidence-based guidelines from ESPGHAN and NASPGHAN for Helicobacter pylori infection in children. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):230-43. doi: 10.1097/MPG.0b013e3182227e90. PMID 21558964
- [Background] Zhou L, Zhang J, Song Z, He L, Li Y, Qian J, Bai P, Xue Y, Wang Y, Lin S. Tailored versus Triple plus Bismuth or Concomitant Therapy as Initial Helicobacter pylori Treatment: A Randomized Trial. Helicobacter. 2016 Apr;21(2):91-9. doi: 10.1111/hel.12242. Epub 2015 Jun 23. PMID 26104022
- [Background] Seo JH, Woo HO, Youn HS, Rhee KH. Antibiotics resistance of Helicobacter pylori and treatment modalities in children with H. pylori infection. Korean J Pediatr. 2014 Feb;57(2):67-71. doi: 10.3345/kjp.2014.57.2.67. Epub 2014 Feb 24. PMID 24678329
- [Background] Homan M, Hojsak I, Kolacek S. Helicobacter pylori in pediatrics. Helicobacter. 2012 Sep;17 Suppl 1:43-8. doi: 10.1111/j.1523-5378.2012.00982.x. PMID 22958155
- [Background] Erdur B, Ozturk Y, Gurbuz ED, Yilmaz O. Comparison of sequential and standard therapy for Helicobacter pylori eradication in children and investigation of clarithromycin resistance. J Pediatr Gastroenterol Nutr. 2012 Nov;55(5):530-3. doi: 10.1097/MPG.0b013e3182575f9c. PMID 22465935 (Retraction: PMID 23325443 Branski D, Heyman MB. J Pediatr Gastroenterol Nutr. 2013 Feb;56(2):239)
- [Background] Bontems P, Kalach N, Oderda G, Salame A, Muyshont L, Miendje DY, Raymond J, Cadranel S, Scaillon M. Sequential therapy versus tailored triple therapies for Helicobacter pylori infection in children. J Pediatr Gastroenterol Nutr. 2011 Dec;53(6):646-50. doi: 10.1097/MPG.0b013e318229c769. PMID 21701406
- [Background] Mehri N, Kambiz E, Ahmad K, Fatemeh F, Farzaneh M, Hossein FG, Fatemeh M. The efficacy of a 1-week triple therapy for eradication of Helicobacter pylori infection in children. Arab J Gastroenterol. 2011 Mar;12(1):37-9. doi: 10.1016/j.ajg.2011.01.011. Epub 2011 Feb 5. PMID 21429454